CLINICAL TRIAL: NCT02425813
Title: Intra-Arterial Steroid Administration of De Novo Acute Graft-vs-Host Disease of the Gastrointestinal Tract: A Phase II Study
Brief Title: Methylprednisolone Sodium Succinate in Treating Patients With Acute Graft-versus-Host Disease of the Gastrointestinal Tract
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00032434; NCI-2015-00548 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98115 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-24 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Acute Graft Versus Host Disease; Intestinal Graft Versus Host Disease
MeSH Terms: interventions — Budesonide; Methylprednisolone Hemisuccinate; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (methylprednisolone sodium succinate, budesonide) (Experimental): STUDY AGENT: Patients receive methylprednisolone sodium succinate IA QD on days 1-3.
  CONVENTIONAL THERAPY: Patients also receive conventional therapy comprising methylprednisolone sodium succinate IV every 12 hours on for 7-14 days beginning on day 1 and budesonide PO on days 1-56. Patients with response by day 7-14 may begin taper and receive methylprednisolone PO on days 28-56. Treatment continues in the absence of disease progression or unacceptable toxicity.
  IST: Patients receive conventional IST or continue their previous prophylactic regimen beginning on day 1 to 56 (or beyond) at the discretion of the treating physician.
  Interventions: Drug: Budesonide; Drug: Methylprednisolone Sodium Succinate

INTERVENTIONS:
Drug: Budesonide — Given PO
  Other Names: Budecort; Butacort; Eltair; Nasocort; Preferid; Pulmicort; Pulmicort Turbuhaler; Rhinocort
Drug: Methylprednisolone Sodium Succinate — Given IA and IV
  Other Names: A-MethaPred; Asmacortone; Cryosolona; Medrate; Metypred; Prednilem; Solu Moderin; Solu-Medrol; Solu-Medrone

SUMMARY:
This phase II trial studies how well methylprednisolone sodium succinate works in treating patients with graft-versus-host disease (GVHD) of the gastrointestinal tract that has begun within 100 days of transplant (acute GVHD). Corticosteroids are a type of drug that reduces inflammation. Giving corticosteroid drugs, such as methylprednisolone sodium succinate, directly into the arteries of the gastrointestinal tract may help treat inflammation caused by GVHD. Giving methylprednisolone sodium succinate in addition to standard treatments may be more effective in treating GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of intra-arterial steroid administration (IASA) with methylprednisolone sodium succinate (MePDSL) in this dose-schedule for treatment of de novo acute moderate-to-severe GvHD of the gastrointestinal tract (GIT).

SECONDARY OBJECTIVES:

I. To assess the safety of IASA MePDSL in this dose-schedule for treatment of de novo acute moderate-to-severe acute GvHD of the GIT.

II. To assess the feasibility of IASA MePDSL in this dose-schedule for treatment of de novo acute moderate-to-severe acute GvHD of the GIT.

OUTLINE:

STUDY AGENT: Patients receive methylprednisolone sodium succinate intra-arterially (IA) once daily (QD) on days 1-3.

CONVENTIONAL THERAPY: Patients also receive conventional therapy comprising methylprednisolone sodium succinate intravenously (IV) every 12 hours on for 7-14 days beginning on day 1 and budesonide PO on days 1-56. Patients with response by day 7-14 may begin taper and receive methylprednisolone orally (PO) on days 28-56. Treatment continues in the absence of disease progression or unacceptable toxicity.

IMMUNOSUPPRESSIVE THERAPY (IST): Patients receive conventional IST or continue their previous prophylactic regimen beginning on day 1 to 56 (or beyond) at the discretion of the treating physician.

After completion of study treatment, patients are followed up for 360 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute GvHD of the GIT (any site except isolated "upper" GIT disease); other sites may be involved as well; their presence will not influence eligibility

  * Biopsies are strongly recommended and should be obtained, ideally, by full endoscopy including esophagogastroduodenoscopy (EGD) and flexible sigmoidoscopy or colonoscopy
  * However, and with an appropriate clinical presentation, it is desirable -- but not necessary -- to have pathology confirmation
  * If other diagnoses are excluded, it is not necessary to biopsy all potentially involved sites in the GIT to initiate therapy
  * It is possible that other diagnoses may be present as well, and this should not exclude eligibility so long as they are distinct (this statement is generic, but applies especially to various types of infective colitis; that said, on-going anti-infective therapy must be on-going)
* Any diagnosis, donor or source of hematopoietic stem cells (HSC) is allowed, including donor leukocyte infusions (DLI)
* Prior or on-going therapy:

  * De novo disease with no previous systemic (topical allowed) therapy for acute GvHD --except for a maximum (and ideally much less) of 72 hours of prior glucocorticoid (GC) therapy, > 0.5 mg/kg/day of MePDSL or equivalent after the onset of acute GvHD
  * An exception to the above exists for patients with prior acute GvHD (of any site) who received GC therapy, experienced a complete response (CR), were tapered off GC and recurred >= 15 days later; such are eligible after review by the principal investigator (PI) or his designee
  * The use of on-going acute GvHD prophylaxis will be continued
  * The use of any other IST is allowed if acute GvHD of the GIT develops while the patient is off all IST; IST may be started at the discretion of the attending physician after discussion with the PI of this study
  * Treatment with oral budesonide is to be started or continued at full dose
  * Please consult with the study PI regarding any questions or concerns of study eligibility
* No specific organ function parameters are required; however, significant abnormalities should be discussed with the study PI
* Ability to understand and the willingness to sign the Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Significant risk factors for IASA therapy including, but not limited to: major uncorrectable coagulopathy, bowel perforation, ongoing bacteremia, mesenteric insufficiency, etc; in these or any questionable cases, discussion with the PI is recommended
* Patients may not be receiving any other drugs for the treatment of GvHD or investigational agents, except for a maximum of 72 hours of prior GC therapy, as above
* Uncontrolled, severe infective processes
* Patients with relapsed or persistent malignancy requiring immunosuppressive withdrawal or modulation (an example of this may be a patient who relapsed and was being treatment with DLI and then developed GvHD)
* Pregnant women are excluded from this study; breastfeeding should be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of discontinuation of systemic GCs without acute GvHD flare and without disease progression/recurrence | Day 56
Incidence of discontinuation of systemic GCs without acute GvHD flare and without disease progression/recurrence | By day 180
Incidence of discontinuation of systemic GCs without acute GvHD flare and without disease progression/recurrence | By day 360
Proportions of response among surviving patients | Day 14
Proportions of progression among surviving patients | Day 14
Rate of acute (and/or chronic) GvHD-free survival | Day 56
  Simon's two-stage design will be used. The null hypothesis that the true CR rate is 30% will be tested against a one-sided alternative and presented with a 95% confidence interval.
Proportions of response among surviving patients | Day 28
Proportions of progression among surviving patients | Day 28

SECONDARY OUTCOMES:
Daily and cumulative GC dose | Day 28
  Descriptive measures will be provided at each time point specified.
Feasibility | Up to day 360
  Feasibility will be defined as less than three IASA sessions for any reason and obvious procedure-related problems in >= 10% of patients. Descriptive measures will be provided at each time point specified.
GvHD-free survival | Day 180
  Descriptive measures will be provided at each time point specified. Survival estimates will be calculated using Kaplan-Meier estimation.
GvHD-free survival | Day 360
  Descriptive measures will be provided at each time point specified. Survival estimates will be calculated using Kaplan-Meier estimation.
Incidence of acute GvHD "flare" after CR/PR requiring modification and/or additional agents (and/or 2.5 mg/kg/day of prednisone [or methylprednisolone equivalent of 2 mg/kg/day]) for systemic therapy | Up to day 56
  Descriptive measures will be provided at each time point specified.
Incidence of chronic GvHD | By day 180
  Descriptive measures will be provided at each time point specified.
Incidence of chronic GvHD | By day 360
  Descriptive measures will be provided at each time point specified.
Incidence of National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 toxicities | Up to day 360
  Frequencies of toxicities grade 2 or higher will be totaled at the conclusion of the study.
Incidence of opportunistic infections | Day 180
  Descriptive measures will be provided at each time point specified.
Non-relapse mortality (NRM) | Day 180
  Descriptive measures will be provided at each time point specified.
NRM | Day 360
  Descriptive measures will be provided at each time point specified.
Overall survival | Day 180
  Descriptive measures will be provided at each time point specified. Survival estimates will be calculated using Kaplan-Meier estimation.
Overall survival | Day 360
  Descriptive measures will be provided at each time point specified. Survival estimates will be calculated using Kaplan-Meier estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Phillips, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States